CLINICAL TRIAL: NCT04582487
Title: Advancing Chemical and Genomic Strategies for Relapsed/Refractory T-ALL and ETP-ALL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ALL2720
Record Dates: First submitted 2020-09-24; First posted 2020-10-09 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: T Acute Lymphoblastic Leukemia; Early T Acute Lymphoblastic Leukemia; T-lymphoblastic Lymphoma; Etp All
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological evaluation (Other): A combined approach of Drug Sensitivity and Resistance Profiling (DSRP) and molecular-cytogenetic findings is used in order to prioritize compounds for tailored therapies.
  Interventions: Other: bone marrow and/or peripheral blood samples withdrawal

INTERVENTIONS:
Other: bone marrow and/or peripheral blood samples withdrawal — bone marrow and/or peripheral blood samples evaluation

SUMMARY:
This is a biological study for R/R T-ALL/LBL or ETP-ALL patients. Bone marrow and/or peripheral blood samples will be subjected to genomic, DSRP profiling and phosphoproteomic screening to identify novel potential therapeutic approach and thus, eligibility for treatment based on molecular and DSRP data. As soon as genomic and DSRP profiling are made available, local Investigator can submit to local ethic committee a request for clinical use of identified compound.

DETAILED DESCRIPTION:
This is a biological study for R/R T-ALL/LBL or ETP-ALL patients. Bone marrow and/or peripheral blood samples will be subjected to genomic, DSRP profiling and phosphoproteomic screening to identify novel potential therapeutic approach and thus, eligibility for treatment based on molecular and DSRP data.

Genomic studies include karyotyping, CI-FISH and sequencing of 72 selected genes recurrently involved in T-ALL (by NGS).

A panel of 80 compounds has been choosen for DSRP profile.

As soon as genomic and DSRP profiling are made available, local Investigator can submit to local ethic committee a request for clinical use of compound hits. Meanwhile, in case of leukocytosis and uncontrolled disease, patients will be treated with cytoreductive therapies and best supportive care according to guidelines and scientific consensus.

Every patient will receive a molecularly and functionally informed therapy following the therapeutic schedule already defined by in other tumors. Treatment will be selected on the basis of integration of genomic and small response data.

ELIGIBILITY:
Inclusion Criteria:

* Patients to be enrolled in this study must have T-cell ALL or T-cell lymphoblastic lymphoma (LL) in the first relapse or must have failed primary induction chemotherapy (i.e., never attained a complete remission following an initial course of standard therapy for T-ALL/LBL or have a diagnosis of ETP-ALL [T-ALL with the following phenotype: Negative: CD1a-, CD8-, CD4-, CD5 (less than 75% of blasts); CD13+, CD33+, CD34+, CD117+, HLA-DR+, CD11b+, and/or CD65+ -in at least 25% of lymphoblasts
* Ages Eligible for Study: over 18 years
* Patients with T-ALL/LBL must have greater than 5% blasts in the bone marrow with or without extramedullary disease
* Patients with T-ALL/LBL must have recurrent disease, documented by clinical or radiographic criteria, as well as histologic verification of the malignancy at original diagnosis
* Patients may have CNS 1 (WBC count in CSF <5 and having no blasts) or CNS 2 (WBC count in CSF <5 and having blasts) disease but not CNS 3 (WBC count in CSF ≥5 and having blasts)
* ECOG 0-2 or Karnofsky ≥ 50%
* Patients may be enrolled on study regardless of the timing of prior Intrathecal therapy; however, they may not begin treatment on this protocol until a minimum of 7 days has elapsed since prior intrathecal therapy
* Adequate renal function defined as serum creatinine ≤ 1.5x upper limit of normal (ULN) for age. If the serum creatinine is above these values, the calculated creatinine clearance or radioisotope GFR must be ≥ 70 mL/min/1.73m2
* Total bilirubin ≤ 1.5x ULN for age. If the total bilirubin is elevated, patient will still be eligible if the conjugated (direct) serum bilirubin ≤ ULN for age
* ALT ≤ 5x ULN of normal for age
* Adequate cardiac function defined as shortening fraction of ≥ 27% by echocardiogram or ejection fraction ≥ 45% by gated radionuclide study
* No evidence of dyspnea at rest
* No exercise intolerance
* A pulse oximetry ≥ 94% at sea level (≥ 90% at altitude ≥ 5000 feet) if there is clinical indication for determination
* Patients must be capable of understanding the investigational nature, potential risks and benefits of the study. All patients must sign a written informed consent

Exclusion Criteria:

* Significant organ compromise that will increase risk of toxicity or mortality
* Active serious infection not controlled by oral or intravenous antibiotics
* Active secondary malignancy other than skin cancer (e.g., basal cell carcinoma or squamous cell carcinoma) that in the investigator's opinion will shorten survival to less than 1 year
* Known hepatitis B or C infection, or known seropositivity for human immunodeficiency virus (HIV)
* Active grade III-V cardiac failure as defined by the New York Heart Association Criteria
* Patients with a cardiac ejection fraction (as measured by either multigated acquisition [MUGA] or echocardiogram) < 40%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-05-19 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Drug sensitivity profile | baseline
  Frequencies of alternative therapies identified for T-ALL patients

CONTACTS AND LOCATIONS:
Locations (10):
- Italy (10):
  - Aou Ospedali Riuniti "Umberto I - G.M. Lancisi - G. Salesi"- Ancona - Sod Clinica Ematologica, Ancona
  - Asst Papa Giovanni Xxiii - Ospedale Di Bergamo - Sc Ematologia, Bergamo
  - Aou Di Bologna - Policlinico S. Orsola-Malpighi - Uoc Ematologia, Bologna
  - Asst Degli Spedali Civili Di Brescia - Uo Ematologia, Brescia
  - Asl Lecce, Ospedale 'V. Fazzi' - Uo Ematologia, Lecce
  - Aulss 3 Serenissima, Ospedale Dell'Angelo - Mestre - Uo Ematologia, Mestre
  - Ematologia ed Immunologia Clinica, Perugia
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs - Roma - Area Ematologica, Roma
  - Aou Senese - Uoc Ematologia E Trapianti, Siena
  - Aulss 8 Berica - Ospedale Di Vicenza - Uoc Ematologia, Vicenza